CLINICAL TRIAL: NCT04180020
Title: Coordinating Opioid Use Treatment Through Medical Management With Infection Treatment (Project COMMIT)
Acronym: COMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000026223; U01TR002763 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAU (Active Comparator): Treatment as Usual (TAU).
  Interventions: Other: TAU
- ID/LAB (Experimental): Infectious Disease management of OUD with Long-Acting injectable buprenorphine (ID/LAB).
  Interventions: Other: ID/LAB

INTERVENTIONS:
Other: ID/LAB — ID/LAB is the new model in which OUD is managed by Infectious Disease (ID) specialists and/or Hospitalists concurrent with management of the infectious diseases, using long-acting injectable buprenorphine (LAB).
  Arms: ID/LAB
Other: TAU — TAU is designed to systematize what is the current practice at the participating hospitals and in most U.S. hospitals while offering a minimum standard of care. TAU will constitute recommendation for MOUD initiation and consultation for addiction medicine when available; in practice, it is typically detoxification from opioids and referral to community-based addiction treatment after hospital discharge.
  Arms: TAU

SUMMARY:
This study seeks to test a new model of care (ID/LAB) in which opioid use disorder (OUD) is managed by infectious disease (ID) specialists and hospitalists concurrent with management of the OUD-related infections, using long-acting injectable buprenorphine (LAB), followed by referral as soon as possible after hospital discharge to community resources for long term treatment of OUD.

DETAILED DESCRIPTION:
There are three specific aims that this study will use to assess a new model of care aimed at treating opioid use disorder (OUD). These aims address whether treatment is maintained by patients, if patients' opioid use outcomes improve and to determine if adherence to treatment for infectious disease results in fewer re-hospitalizations and emergency room visits, as well as improved quality of life.

The specific aims:

Aim1: The primary outcome will be a binary indicator of whether a patient is enrolled in and receiving effective medication treatment for OUD (buprenorphine, methadone, or injection naltrexone) at 12 weeks (3 months) after randomization.

Aim 2: Evidence of improved opioid use outcomes (lower days of using opioids, negative urine opioids).

Aim 3: Have higher rates of completion of the antimicrobial regimen for their infectious disease, decreased re-hospitalizations and emergency room presentations related to either their infectious disease or OUD over the 12-week follow-up period, and improved measures of quality of life.

The intent of this study is to test the hypothesis:

Assignment to the ID/LAB arm (OUD managed directly by the infectious disease (ID) specialists or hospitalist team with long acting injection buprenorphine (LAB)) will promote greater enrollment in effective medication treatment for OUD at 12 weeks after randomization, compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

* Adults able to provide written informed consent in English or Spanish;
* Current hospitalization with a suspected or known bacterial or viral (HIV/HCV/HBV) infection including but not limited to bacteremia, Candidal fungemia, osteomyelitis, endophthalmitis, septic thrombophlebitis, infected pseudoaneurysm, endocarditis, skin/soft tissue infection (SSTI), or septic arthritis;
* Current moderate-to-severe OUD (DSM-5);
* Willing to accept assignment to either ID/LAB or TAU, and to participate in research follow-up visits.

Exclusion Criteria:

* Severe medical or psychiatric disability making participation unsafe (e.g. imminent suicide risk);
* Pregnancy, planning conception, or breast-feeding for female participants;
* Allergy, hypersensitivity or medical contraindication to buprenorphine;
* Moderate-severe liver impairment in the judgment of the study investigator;
* Preexisting enrollment on methadone or buprenorphine (SL-B) maintenance AND intending to remain on methadone or buprenorphine maintenance upon discharge (patients already under effective treatment for OUD do not represent the target population of untreated OUD patients entering hospitals, nor would we want to disrupt established effective treatment).
* Inability or unwillingness of subject to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Springer, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Prisma Health, Greenville, South Carolina

REFERENCES:
- [Derived] Seval N, Roth P, Frank CA, Di Paola A, Litwin AH, Vander Wyk B, Neirinckx V, Schlossberg E, Lawson P, Strong M, Schade MA, Nunez J, Levin FR, Brady KT, Nunes EV, Springer SA. Initiating Injectable Buprenorphine in People Hospitalized With Infections: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2513000. doi: 10.1001/jamanetworkopen.2025.13000. PMID 40445619

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual (TAU).: Treatment as Usual (TAU).
  TAU: TAU is designed to systematize what is the current practice at the participating hospitals and in most U.S. hospitals while offering a minimum standard of care. TAU will constitute recommendation for MOUD initiation and consultation for addiction medicine when available; in practice, it is typically detoxification from opioids and referral to community-based addiction treatment after hospital discharge.
Period: Overall Study
Arm/Group | Treatment as Usual (TAU). | ID/LAB
Started | 85 | 86
Missed 12 Week Visit | 18 | 16
Completed (completed 12 week visit) | 63 | 59
Not Completed | 22 | 27
Not completed — missed visit | 18 | 16
Not completed — Death | 2 | 3
Not completed — Withdrawal by Subject | 1 | 5
Not completed — incarcerated | 1 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU). | ID/LAB | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [33 to 47] | 38 [32 to 46] | 39 [33 to 47]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men | 42 | 46 | 88
  Women | 43 | 39 | 82
  Transgender women | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 4 | 18
  Not Hispanic or Latino | 71 | 82 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 63 | 74 | 137
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 85 | 86 | 171
Housing Status [Count of Participants; unit: Participants]
  Unhoused | 21 | 21 | 42
  Unstable Housing | 37 | 30 | 67
  Stable Housing | 27 | 34 | 61
  Unknown or Not Reported | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  High School or above | 68 | 67 | 135
  Less than high school | 17 | 17 | 34
  Did not respond | 0 | 2 | 2
Marital Status [Count of Participants; unit: Participants]
  Living with partner | 5 | 12 | 17
  Married | 10 | 11 | 21
  Divorced | 18 | 21 | 39
  Never married | 40 | 29 | 69
  Separated | 10 | 8 | 18
  Widowed | 2 | 4 | 6
  Unknown or Not Reported | 0 | 1 | 1
Income group [Count of Participants; unit: Participants]
  Less than $5,000 | 27 | 25 | 52
  $5,000-9,999 | 6 | 6 | 12
  $10.000-24,999 | 20 | 16 | 36
  $25,000-49,999 | 16 | 17 | 33
  $50,000 or more | 15 | 17 | 32
  Unknown or Not Reported | 1 | 5 | 6
Type of insurance [Count of Participants; unit: Participants]
  Medicaid | 38 | 38 | 76
  Medicare | 1 | 2 | 3
  Private insurance | 6 | 7 | 13
  Other insurance | 1 | 3 | 4
  None | 39 | 35 | 74
  Did not respond | 0 | 1 | 1
Engaged in condomless sex [Count of Participants; unit: Participants]
  Yes | 48 | 46 | 94
  No | 36 | 35 | 71
  Did not respond | 1 | 5 | 6
Median number of condomless sex partners [Median (Inter-Quartile Range); unit: partners] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
WHO Quality of Life-BREF (WHOQOL-BREF) [Median (Inter-Quartile Range); unit: score on a scale] — Assesses quality of life in four domains: physical health, psychological, social relationships and environment. The domain scores were transformed into a linear scale with a range of 0-100. Higher scores indicate a better quality of life.
  score on a scale
    Physical Health | 42.9 [28.6 to 60.7] | 39.3 [21.4 to 57.1] | 39.3 [25.5 to 60.7]
    Psychological | 45.8 [37.5 to 62.5] | 45.8 [37.5 to 66.7] | 45.8 [37.5 to 62.5]
    Social Relationships | 45.8 [29.2 to 66.7] | 54.2 [29.2 to 75.0] | 50.0 [29.2 to 75]
    Environmental | 53.1 [40.6 to 68.8] | 56.7 [40.6 to 78.1] | 56.3 [40.6 to 71.9]
Provisional Post-traumatic stress disorder (PTSD) Diagnosis [Count of Participants; unit: Participants] — Diagnosed via the Post-Traumatic Diagnostic Scale 5 (PTSD - PCL)
  Participants | 48 | 45 | 93
Depression Severity [Count of Participants; unit: Participants] — Diagnosed via Patient Health Questionnaire-9 (PHQ-9)
  Participants
    None or mild | 26 | 23 | 49
    Moderate or above | 57 | 60 | 117
    Did not answer | 2 | 3 | 5
Provisional Attention-deficit/hyperactivity disorder (ADHD) [Count of Participants; unit: Participants] — Diagnosed via Adult ADHD Self-Report Scale
  Participants | 50 | 62 | 112
Pain Scale score via Pain, Enjoyment of Life and General Activity (PEG) Scale [Median (Inter-Quartile Range); unit: score on a scale] — Scored on a scale of 0-10. A higher score indicates more pain and worse functioning.
  score on a scale | 6.0 [3.0 to 8.0] | 6.0 [4.0 to 7.0] | 6.0 [3.2 to 7.8]
Opioid Craving Scale [Median (Inter-Quartile Range); unit: score on a scale] — Score range 0-5. Higher scores indicate more cravings.
  score on a scale | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 5.00]
Opioid withdrawal (mild or greater) [Count of Participants; unit: Participants] — Assessed via Clinical Opiate Withdrawal Scale (COWS).
  Participants | 19 | 8 | 27
Hazardous/Harmful Drinking [Count of Participants; unit: Participants] — Assessed via Alcohol Use Disorders Identification Test (AUDIT).
  Participants | 23 | 15 | 38
Co-occurring stimulant use disorder [Count of Participants; unit: Participants] — Assessed via Mini Internation Neuropsychiatric Interview (MINI)
  Participants | 48 | 44 | 92
Prescribed MOUD in past 30 days [Count of Participants; unit: Participants] | 15 | 19 | 34
Positive urine toxicology screen at time of enrollment [Count of Participants; unit: Participants]
  Opiates: Negative | 71 | 61 | 132
  Opiates: Positive | 11 | 23 | 34
  Opiates: Missing | 3 | 2 | 5
  Oxycodone: Negative | 62 | 64 | 126
  Oxycodone: Positive | 20 | 20 | 40
  Oxycodone: Missing | 3 | 2 | 5
  Fentanyl: Negative | 42 | 44 | 86
  Fentanyl: Positive | 39 | 40 | 79
  Fentanyl: Missing | 4 | 2 | 6
  Methadone: Negative | 67 | 62 | 129
  Methadone: Positive | 14 | 22 | 36
  Methadone: Missing | 4 | 2 | 6
  Buprenorphine: Negative | 29 | 27 | 56
  Buprenorphine: Positive | 51 | 57 | 108
  Buprenorphine: Missing | 5 | 2 | 7
  Cocaine: Negative | 77 | 81 | 158
  Cocaine: Positive | 5 | 3 | 8
  Cocaine: Missing | 3 | 2 | 5
  Methamphetamine: Negative | 70 | 77 | 147
  Methamphetamine: Positive | 12 | 7 | 19
  Methamphetamine: Missing | 3 | 2 | 5
  Benzodiazepine: Negative | 62 | 55 | 117
  Benzodiazepine: Positive | 20 | 29 | 49
  Benzodiazepine: Missing | 3 | 2 | 5
Self-reported substances used 30 days prior to hospitalization [Count of Participants; unit: Participants] — Assessed via TLFB
  Participants
    Heroin: No | 27 | 27 | 54
    Heroin: Yes | 57 | 58 | 115
    Heroin: Missing | 1 | 1 | 2
    Prescription opioids: No | 68 | 64 | 132
    Prescription opioids: Yes | 16 | 21 | 37
    Prescription opioids: Missing | 1 | 1 | 2
    Fentanyl: No | 45 | 49 | 94
    Fentanyl: Yes | 39 | 36 | 75
    Fentanyl: Missing | 1 | 1 | 2
    Other opioids: No | 78 | 76 | 154
    Other opioids: Yes | 6 | 9 | 15
    Other opioids: Missing | 1 | 1 | 2
    Cocaine: No | 56 | 55 | 111
    Cocaine: Yes | 28 | 30 | 58
    Cocaine: Missing | 1 | 1 | 2
    Methamphetamine: No | 45 | 44 | 89
    Methamphetamine: Yes | 39 | 41 | 80
    Methamphetamine: Missing | 1 | 1 | 2
Visited health care provider in last 12 months, excluding urgent care [Count of Participants; unit: Participants] | 34 | 28 | 62
Covered by health insurance 30 days before interview [Count of Participants; unit: Participants] | 46 | 50 | 96
Engaged in injection drug use [Count of Participants; unit: Participants]
  No | 31 | 21 | 52
  Yes | 53 | 64 | 117
  Missing | 1 | 1 | 2
Shared injection drug equipment [Count of Participants; unit: Participants]
  No | 35 | 42 | 77
  Yes | 18 | 21 | 39
  Missing | 1 | 2 | 3
  Does not apply | 31 | 21 | 52
Index Infection [Count of Participants; unit: Participants]
  HIV diagnosis | 3 | 1 | 4
  HIV viral load ≥ 200 | 0 | 1 | 1
  Hepatitis C, Ab positive | 53 | 61 | 114
  Hepatitis C, with detectable viral load | 36 | 35 | 71
  Hepatitis B | 0 | 2 | 2
  Bloodstream infection | 36 | 41 | 77
  Endocarditis | 15 | 20 | 35
  Septic arthritis | 14 | 14 | 28
  Osteomyelitis | 16 | 15 | 31
  Pneumonia/respiratory infection (non-COVID-19) | 19 | 14 | 33
  Septic thrombophlebitis | 2 | 2 | 4
  Skin/skin structure infection | 11 | 24 | 35
  Abscess including skin/soft tissue, intra-abdominal, epidural, and other | 30 | 27 | 57
  COVID-19 Infection | 3 | 3 | 6
  Sexually transmitted infection | 3 | 5 | 8
  Other | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Retention in Medication Treatment for OUD
Description: Enrollment in effective medication treatment for OUD (either buprenorphine maintenance, methadone maintenance, or extended-release naltrexone) will be ascertained through interview of the participant at each assessment point, using a modified, brief version of the Treatment Services Review that records type and dose of medication treatment, contact information on the treatment program, and psychosocial treatment modalities accessed since the previous visit (e.g. professional counseling, 12-step group participation).
  The primary outcome will be a binary indicator of whether or not the patient is enrolled on buprenorphine maintenance treatment or other effective medication (methadone maintenance or extended-release naltrexone) at 12 weeks after randomization, verified by either report from the treatment program, or if the treatment program does not respond, prescription drug monitoring report or EMR.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU). | ID/LAB
Number analyzed (Participants) | 85 | 86
Participants | 46 | 51
Statistical Analysis 1: Comparison: Treatment as Usual (TAU). vs ID/LAB; Test type: Superiority; p = 0.94, t-test, 2 sided

2. Secondary Outcome: Total Days of Using Opioids
Description: This outcome will be measured by Timeline Followback, which assesses self-reported alcohol and other drug use including opioid use route of use and form of drug, for the 30 days before baseline, and for each day over the follow up period, using calendars and memory aids to enhance recall.
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Total Days of Using Opioids
Description: as for outcome 2
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Total Days of Using Opioids
Description: as for outcome 2
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Total Days of Using Opioids
Description: as for outcome 2
Time Frame: 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Negative Urine Screens: Opioids
Description: This outcome will be measured by urine toxicology-confirmed abstinence via urine toxicology (Manufacturer: Redwood Toxicology) for recent illicit opioid use.
Time Frame: 4 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Negative Urine Screens: Opioids
Description: as for outcome 6
Time Frame: 8 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Negative Urine Screens: Opioids
Description: as for outcome 6
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Negative Urine Screens: Opioids
Description: as for outcome 6
Time Frame: 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Treatment Completion Rate
Description: This outcome is assessed by the Medical/Infectious Disease/TAU questionnaire. This form documents the completion of antimicrobial therapy and re-hospitalization for infection. The initial evaluation documents the relevant infection and medical details such as infection site, organism, and stage. It also extracts the type of ant-infective, route of administration, dose, and planned duration. Information on follow-up is collected alteration of treatment plan, infection related adverse events (e.g. PICC complications, drug reaction/toxicity to anti-infective agent prescribed by non-study clinicians, etc), and intervening hospitalizations. Completion success is defined as appropriate completion of antimicrobial therapy, as documented in the initial assessment, without interruption or unexpected prolongation of therapy.
Time Frame: 4 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Treatment Completion Rate
Description: as for outcome 10
Time Frame: 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Treatment Completion Rate
Description: as for outcome 10
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Treatment Completion Rate
Description: as for outcome 10
Time Frame: 24 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Re-hospitalization/Emergency Room Visits
Description: Re-hospitalizations and emergency room presentations related to either their infectious disease or OUD will be totaled over the intervention duration and 12-week follow-up period.
Time Frame: 12 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Re-hospitalization/Emergency Room Visits
Description: as for outcome 14
Time Frame: 24 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Quality of Life Measure of Social and Occupational Functioning
Description: Quality of life is measured using the WHOQOL-Bref, which is a is a well validated and widely used scale for persons with substance use disorders that measures the quality of social and occupational functioning as well as other domains. Scores are scaled in a positive direction (higher scores indicate a higher quality of life). A total of 500 is the highest score attainable and indicates highest quality of life in respondents.
Time Frame: 12 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Quality of Life Measure of Social and Occupational Functioning
Description: as for outcome 16
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Treatment as Usual (TAU). | ID/LAB
All-Cause Mortality (participants affected / at risk) | 4/85 | 4/86
Serious Adverse Events (participants affected / at risk) | 20/85 | 31/86
Other Adverse Events (participants affected / at risk) | 68/85 | 67/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment as Usual (TAU). (N=85) | ID/LAB (N=86)
Opioid Withdrawal (Nervous system disorders) | 1 | 0
Skin/soft tissue infection (Skin and subcutaneous tissue disorders) | 14 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-fatal opioid overdose (Nervous system disorders) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Respiratory infection (not including COVID-19) (Infections and infestations) | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment as Usual (TAU). (N=85) | ID/LAB (N=86)
Opioid Withdrawal (Nervous system disorders) | 9 | 14
Skin/soft tissue infection (Skin and subcutaneous tissue disorders) | 9 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8
Nausea (Gastrointestinal disorders) | 5 | 10
Rash (Skin and subcutaneous tissue disorders) | 7 | 7
Headache (Nervous system disorders) | 4 | 9
Edema (Vascular disorders) | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Injection site reaction (General disorders) | 0 | 9
Vomiting (Gastrointestinal disorders) | 4 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 1 | 7
Diaphoresis (General disorders) | 3 | 4
Fatigue (General disorders) | 5 | 2
Fever (Immune system disorders) | 3 | 4
Non-fatal opioid overdose (Nervous system disorders) | 6 | 1
Insomnia (Nervous system disorders) | 2 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Respiratory infection (not including COVID-19) (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04180020/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04180020/ICF_001.pdf